CLINICAL TRIAL: NCT02580344
Title: Action of Ibuprofen on IUD-associated Heavy Menstrual Bleeding
Brief Title: The Effect of Ibuprofen on Intrauterine Contraceptive Device Associated Uterine Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUD_Ibuprofen
Record Dates: First submitted 2015-10-18; First posted 2015-10-20 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Contraception
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibuprofen (Other)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — The women will receive 400mg ibuprofen 3 times per day from the first day of the cycle for 5 days

SUMMARY:
The Copper intrauterine device is the most common method of reversible contraception worldwide. Abnormal uterine bleeding and pain are the most common medical indications for the discontinuation of the intrauterine device.

Excessive prostaglandin release in the endometrial cavity appears to play an important role in both bleeding and pain related to copper intrauterine devices.There are many types of prostaglandin metabolites that present in the endometrium one of them is prostacyclin which causes vasodilatation and inhibits platelet aggregation. Another one is thromboxane which has two types; A2 which is active and rapidly converted into B2, which is inactive. Thromboxane causes vasoconstriction and blood clotting.

Non-steroidal anti-inflammatory drugs (NSAIDs) are prostaglandin synthetase inhibitors acting by decreasing production of endometrial prostaglandins; they can improve both heavy uterine bleeding and pain. Since its discovery; several drugs in NSAIDs class have been used to treat heavy uterine bleeding and pain associated with copper intrauterine device use such as mefenamic acid, ibuprofen and naproxen.

The most recent systematic review found NSAIDs is the most widely studied drugs for reduction of the menstrual blood and pain associated with copper intrauterine device. The Cochrane Review also found that NSAIDs are the most effective treatment to reduce the bleeding with copper intrauterine device use.

ELIGIBILITY:
Inclusion Criteria:

1. Women have menorrhagia secondary to IUD.
2. Planning for birth spacing for at least 1 year.
3. Patient aged between 20-45 years old.
4. No history of any medical treatment.
5. Living in a nearby area to make follow-up reasonably possible.

Exclusion Criteria:

1. Evidence of defective coagulation.
2. History or evidence of malignancy.
3. Hyperplasia in the endometrial biopsy.
4. Incidental adnexal abnormality on ultrasound.
5. Untreated abnormal cervical cytology
6. contraindications to ibuprofen

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of bleeding days per month | 3 months
  by menstrual diary

SECONDARY OUTCOMES:
Uterine Doppler indices | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes